CLINICAL TRIAL: NCT06401031
Title: The Effect of Auricular Press Needle on Visual Analogue Scale (VAS) and Short Form (SF-12) Scores in Chronic Pain With Depression Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fransisca Pekerti, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-04-0571
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Depressive Symptoms
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Press Needle (Experimental): Device: Press Needle Press needle is a very small needles (1-3 mm long) that are 'pressed' onto acupuncture point and are held in place with a small, sterile surgical adhesive patch.
  Interventions: Device: Press Needle
- Sham Comparator: Sham Press Needle (Sham Comparator): Device: Sham Press Needle Sham press needle is a surgical adhesive patch placed on acupuncture points
  Interventions: Device: Sham Press Needle

INTERVENTIONS:
Device: Press Needle — Press needle is patch-type acupuncture needle which has a very small needle. This is placed onto acupuncture point and give a simultaneous stimulation, which is held in place with a small, sterile surgical adhesive patch.
  Arms: Experimental: Press Needle
Device: Sham Press Needle — Sham press needle is a surgical adhesive patch without needle, that is placed onto acupuncture point
  Arms: Sham Comparator: Sham Press Needle

SUMMARY:
Chronic pain is a medical and social problem that can significantly impact the quality of life. Chronic pain is an important risk factor in the development of depression. It is shown by the significantly higher prevalence of depression in individuals who experience chronic pain (20-80%). Apart from that, chronic pain and depression also have a close relationship in the development of disease and mutually influence the severity of each condition.

To reduce the cost of pain management from a pharmacological perspective and its use in the long term, it is necessary to consider other non-pharmacological treatment methods that have good therapeutic effects with minimal side effects. Acupuncture has become a non-pharmacological therapy option that has proven its effectiveness and safety in treating chronic pain in depressed patients. Previous literature has reported the effectiveness of acupuncture therapy, especially auricular acupuncture in treating pain. Auricular acupuncture therapy using press needles is quite easy to apply, fast, and can provide continuous stimulation with minimal side effects.

This study aimed to assess the effectiveness of the auricular needle press in chronic pain with depressive symptoms. This study was a double-blinded randomized clinical trial and was carried out on outpatients at Dr. Cipto Mangunkusumo National General Hospital Jakarta and Soerojo Hospital Magelang. This is also a collaborative study between the medical acupuncture department and the psychiatry department.

This study includes 60 participants who will be randomly allocated into 2 groups, the press needle and sham press needle groups. The press needles will be placed at 6 auricular points bilaterally, which are MA-TF1 Shenmen, MA-IC7 Heart, and MA-IT1 Cingulate gyrus.

The outcomes that will be assessed in this study are pain intensity using the visual analog scale (VAS) and quality of life using the short form-12 (SF-12) as well as time-to-event achievement in the form of a decrease in the VAS score >= 14 mm.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-59 years.
* Subjects who experience chronic pain with symptoms of depression.
* Subjects with VAS >= 30 mm and < 70 mm from 100 mm during activity (daily activities or light exercise).
* Duration of pain > 3 months.
* Patient Health Questionnaire-9 Items (PHQ-9) score 5-19 on a scale of 0-27.
* Willing to take part in this study until completion and sign the informed consent.

Exclusion Criteria:

* Pain caused by malignancy.
* Patients diagnosed with major depression, depressive symptoms accompanied by psychotic symptoms, and depressive symptoms with antidepressant therapy.
* Patients with medical emergencies or pregnancy.
* Infection, scar tissue, or malignancy at the acupuncture area.
* Anatomical abnormalities in the ear shape.
* Having hypersensitivity reaction to previous acupuncture therapy (metal allergy, atopy, keloid, or other skin hypersensitivity).
* Patients with cognitive impairment or impaired consciousness.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | [Time Frame: first 24 hours, the third day, seventh day, and fourteenth-day post intervention]
  The visual analog scale is measured using a visual ruler with a line scale of 10 cm, where patients are asked to draw a line on the ruler according to the pain they are experiencing. The minimum score is 0 which indicates no pain and the maximum score is 10 which indicates the worst pain. Pain scale measurements are taken every hour in the first 24 hours, on the third day, seventh day, and fourteenth day where a lower scale indicates better progress, which indicates less pain.
Short Form-12 | [Time Frame: on the seventh day and fourteenth-day post-intervention]
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure. The SF-12 is a shortened version of its predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. With a scale from 0 to 100, the scoring yields two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), with a mean of 50 and a standard deviation of 10 in the general population. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.

SECONDARY OUTCOMES:
Time to event | [Time frame: every hour in the first 24 hours post intervention]
  The time to achieve a decrease in the VAS score >= 14 mm (in hours) within the maximum observation period is 24 hours. With a scale 1 to 24 hours, where a lower score indicates better progress, and higher score indicates worse progress.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee ofFaculty of Medicine Universitas Indonesia - RSCM
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No